CLINICAL TRIAL: NCT01740388
Title: A Study to Evaluate the Clinical and Microbial Efficacy of Besifloxacin Ophthalmic Suspension, 0.6% BID Compared to Vehicle in the Treatment of Bacterial Conjunctivitis
Brief Title: Clinical and Microbial Efficacy of Besifloxacin Ophthalmic Suspension, 0.6% in the Treatment of Bacterial Conjunctivitis
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Strategic business decision
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 801
Record Dates: First submitted 2012-11-29; First posted 2012-12-04 (Estimated); Results first posted 2014-09-17 (Estimated); Last update posted 2014-10-01 (Estimated); Status verified 2014-09

CONDITIONS: Bacterial Conjunctivitis
MeSH Terms: conditions — Conjunctivitis, Bacterial | interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Besifloxacin (Experimental): besifloxacin ophthalmic suspension 0.6% administered 2 times daily (BID) for 3 days to participants with a clinical diagnosis of bacterial conjunctivitis
  Interventions: Drug: Besifloxacin
- Vehicle (Placebo Comparator): vehicle of besifloxacin ophthalmic suspension administered 2 times daily (BID) for 3 days to participants with a clinical diagnosis of bacterial conjunctivitis
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Besifloxacin — one drop of besifloxacin ophthalmic suspension 0.6% administered to infected study eye(s) BID for 3 days.
  Other Names: Besivance
  Arms: Besifloxacin
Drug: Vehicle — one drop of the vehicle of besifloxacin ophthalmic suspension administered to infected study eye(s) BID for 3 days.
  Arms: Vehicle

SUMMARY:
To evaluate the clinical and microbial efficacy of besifloxacin ophthalmic suspension, 0.6% (Besifloxacin) administered BID for 3 days compared to vehicle in the treatment of bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Have a clinical diagnosis of acute bacterial conjunctivitis and exhibit mucopurulent/purulent conjunctival discharge (crusty or sticky eyelids) and redness in at least 1 eye. A minimum score of 1 should be present for both discharge and for bulbar conjunctival injection.
* Have monocular pin-holed Snellen visual acuity (VA) equal to or better than 20/200 in both eyes. Age appropriate VA testing will be performed. Every effort should be made to obtain a VA measurement in children. If VA is unobtainable in children, it is at the Investigator's discretion to include the subject in the study.
* Be willing to discontinue contact lens wear for the duration of the study.

Exclusion Criteria:

* Have a severe/serious ocular condition or history/presence of chronic generalized systemic disease that the Investigator feels might increase the risk to the subject or confound the result(s) of the study.
* Have a known hypersensitivity or contraindications to besifloxacin, fluoroquinolones, or any of the ingredients in the study drugs.
* Be expected to require treatment with systemic or ocular (either eye) nonsteroidal anti-inflammatory drugs (NSAIDs), antihistamines, or corticosteroids during the study or have used any of these medications within 2 days prior to study start.
* Be expected to require concurrent ocular therapy in either eye with any ophthalmic solutions (unless specified below), including tear substitutes, during the study or have used any ophthalmic solutions within 2 hours prior to study start. Be expected to require concurrent ocular therapy (either eye) with mast cell stabilizers or decongestants during the study or have used any of the above within 2 days prior to study start.
* Be expected to require concurrent systemic or ocular therapy with immunosuppressants (eg, Restasis) during the study or have used systemic or ocular immunosuppressants within 30 days prior to study start.
* Be expected to require treatment with systemic or ocular (either eye) antibacterials (other than study drug) during the study or have used any systemic or ocular antibacterial within 3 days prior to study start.
* Be likely to require antimicrobial therapy for conditions such as respiratory tract infection, urinary tract infection, skin/soft tissue infection, or otitis media during the study.
* Have had ocular surgery (including laser surgery) in either eye within 6 weeks prior to entry into this study.
* Have suspected viral or allergic conjunctivitis or any other disease conditions that could interfere with the efficacy and safety evaluations of the study medication.
* Have suspected iritis
* Have a history of recurrent corneal erosion syndrome, either idiopathic or secondary to previous corneal trauma or dry eye syndrome.
* Have any active ulcerative keratitis, specifically any epithelial loss greater than punctate keratitis.
* Be immune compromised.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 136 (Actual)
Dates: Start 2013-02; Primary Completion 2013-07 (Actual); Study Completion 2013-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Johnson Varughese, Study Director — Valeant Pharmaceuticals/Bausch & Lomb Incorporated
Locations (1):
- Bausch & Lomb Incorporated, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Besifloxacin | Vehicle
Started | 64 | 72
Completed | 18 | 28
Not Completed | 46 | 44
Not completed — Withdrawal by Subject | 1 | 2
Not completed — Lost to Follow-up | 2 | 0
Not completed — Physician Decision | 2 | 6
Not completed — Subjects missing data, completed | 41 | 36

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Besifloxacin | Vehicle | Total
Number analyzed (Participants) | 64 | 72 | 136
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.6 (22.52) | 50.6 (21.36) | 47.8 (22.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44 | 44 | 88
  Male | 20 | 28 | 48
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 4 | 7 | 11
  Native Hawaiian or Other Pacific Islander | 1 | 1 | 2
  Black or African American | 4 | 7 | 11
  White | 51 | 56 | 107
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 1 | 5

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution
Description: Absence of both conjunctival discharge and bulbar conjunctival injection, after 3 days of treatment with besifloxacin ophthalmic suspension 0.6%
Time Frame: Visit 2 (Day 4 or 5)
Population: Analysis population is only Subjects with non-missing data, Clinical Resolution (LOCF [Last Observation Carried Forward])
Measure: Number; unit: participants
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 18 | 28
participants
  YES | 4 | 5
  NO | 14 | 23

2. Primary Outcome: Microbial Eradication
Description: Absence of all accepted ocular bacterial species that were present at or above threshold at baseline, after 3 days of treatment with besifloxacin ophthalmic suspension 0.6%
Time Frame: Visit 2 (Day 4 or 5)
Population: Analysis population is only Subjects with non-missing data, Microbial Eradication (LOCF [Last Observation Carried Forward])
Measure: Number; unit: participants
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 18 | 28
participants
  YES | 17 | 13
  NO | 1 | 15

3. Secondary Outcome: Clinical Resolution
Description: as for outcome 1
Time Frame: Visit 3 (Day 6, 7, or 8)
Population: as for outcome 1
Measure: Number; unit: participants
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 18 | 28
participants
  YES | 6 | 13
  NO | 12 | 15

4. Secondary Outcome: Microbial Eradication
Description: as for outcome 2
Time Frame: Visit 3 (Day 6, 7, or 8)
Measure: Number; unit: participants
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 18 | 28
participants
  YES | 14 | 16
  NO | 4 | 12

5. Other Pre Specified Outcome: Ocular Conjunctival Discharge
Description: Ocular conjunctival discharge measures on a scale of 0-3 where 0 = Absent, 1 = Mild, 2 = Moderate and 3 = Severe
Time Frame: At each follow-up visit (Visit 1, Visit 2 and Visit 3)
Population: Analysis population is only Subjects with non-missing data, Ocular Discharge Evaluated on the Baseline-Designated Study Eye
Measure: Number; unit: participants
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 18 | 28
participants
  Visit 1: Absent | 0 | 0
  Visit 1: Mild | 6 | 9
  Visit 1: Moderate | 10 | 16
  Visit 1: Severe | 2 | 3
  Visit 2: Absent | 9 | 10
  Visit 2: Mild | 8 | 15
  Visit 2: Moderate | 1 | 2
  Visit 2: Severe | 0 | 0
  Visit 3: Absent | 14 | 16
  Visit 3: Mild | 4 | 5
  Visit 3: Moderate | 0 | 3
  Visit 3: Severe | 0 | 0

6. Other Pre Specified Outcome: Bulbar Conjunctival Injection
Description: Bulbar conjunctival injection measured on a scale of 0-3 where 0 = Normal, 1 = Mild, 2 = Moderate and 3 = Severe
Time Frame: At each follow-up visit (Visit 1, Visit 2 and Visit 3)
Measure: Number; unit: participants
Arm/Group | Besifloxacin | Vehicle
Number analyzed (Participants) | 18 | 28
participants
  Visit 1: Normal | 0 | 0
  Visit 1: Mild | 3 | 6
  Visit 1: Moderate | 14 | 18
  Visit 1: Severe | 1 | 4
  Visit 2: Normal | 4 | 7
  Visit 2: Mild | 13 | 12
  Visit 2: Moderate | 1 | 8
  Visit 2: Severe | 0 | 0
  Visit 3: Normal | 7 | 12
  Visit 3: Mild | 11 | 6
  Visit 3: Moderate | 0 | 5
  Visit 3: Severe | 0 | 1

ADVERSE EVENTS:
Arm/Group | Besifloxacin | Vehicle
Serious Adverse Events (participants affected / at risk) | 0/64 | 0/72
Other Adverse Events (participants affected / at risk) | 2/64 | 3/72
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Besifloxacin (N=64) | Vehicle (N=72)
Conjunctivitis (Eye disorders) | 2 (2) | 1 (1) — Fellow Eye
Eye Pain (Eye disorders) | 0 (0) | 2 (2) — Treated Eye

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less